CLINICAL TRIAL: NCT04160741
Title: Effects of Solar Radiation on Human Function and Cognition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Petros Dinas (Other)
Responsible Party: Sponsor-Investigator, Petros Dinas, Senior Researcher in human physiology, University of Thessaly
Organization: University of Thessaly (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 6. Solar radiation & Thermo
Record Dates: First submitted 2019-11-07; First posted 2019-11-13 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Heat Stress; Heat Strain
Keywords: heat stress; heat strain; solar radiation; responses; cognition; thermal
MeSH Terms: conditions — Heat Stress Disorders | interventions — Radiation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Hot environment with radiation (Experimental): Exposure to hot environment (30°C WBGT) with radiation (800 W/m2)
  Exposure for 03:20:00:
  * rest (two hours)
  * work (cycling) at 100 W (one hour)
  * recovery (twenty minutes)
  Interventions: Other: Radiation and warm environment
- Hot environment without radiation (Experimental): Exposure to hot environment (30°C WBGT) with radiation (0 W/m2)
  Exposure for 03:20:00:
  * rest (two hours)
  * work (cycling) at 100 W (one hour)
  * recovery (twenty minutes)
  Interventions: Other: Warm environment
- Neutral environment with radiation (Experimental): Exposure to neutral environment (20°C WBGT) with radiation (800 W/m2)
  Exposure for 03:20:00:
  * rest (two hours)
  * work (cycling) at 100 W (one hour)
  * recovery (twenty minutes)
  Interventions: Radiation: Neutral environment with radiation
- Neutral environment without radiation (Active Comparator): Exposure to neutral environment (20°C WBGT) with radiation (0 W/m2)
  Exposure for 03:20:00:
  * rest (two hours)
  * work (cycling) at 100 W (one hour)
  * recovery (twenty minutes)
  Interventions: Other: Neutral environment without radiation

INTERVENTIONS:
Other: Radiation and warm environment — Exposure to hot environment (30°C WBGT) with radiation (800 W/m2)
  Exposure for 03:20:00:
  * rest (two hours)
  * work (cycling) at 100 W (one hour)
  * recovery (twenty minutes)
  Arms: Hot environment with radiation
Other: Warm environment — Exposure to hot environment (30°C WBGT) with radiation (0 W/m2)
  Exposure for 03:20:00:
  * rest (two hours)
  * work (cycling) at 100 W (one hour)
  * recovery (twenty minutes)
  Arms: Hot environment without radiation
Radiation: Neutral environment with radiation — Exposure to neutral environment (20°C WBGT) with radiation (800 W/m2)
  Exposure for 03:20:00:
  * rest (two hours)
  * work (cycling) at 100 W (one hour)
  * recovery (twenty minutes)
  Arms: Neutral environment with radiation
Other: Neutral environment without radiation — Exposure to neutral environment (20°C WBGT) with radiation (0 W/m2)
  Exposure for 03:20:00:
  * rest (two hours)
  * work (cycling) at 100 W (one hour)
  * recovery (twenty minutes)
  Arms: Neutral environment without radiation

SUMMARY:
Solar radiation is a physical phenomenon which interacts with any human being throughout its life on earth. This interaction is associated with numerous physiological functions, as well as a broad spectrum of deleterious effects on human health and wellbeing. The aim of this study is to elucidate the effects of solar radiation on human function and cognition in environmental conditions characterized by the same thermal stress.

DETAILED DESCRIPTION:
Volunteers were exposed to four different environmental conditions [two hot environments: 30°C WBGT (1st: air temperature = 32.6°C; relative humidity = 30%; wind speed = 0.5 m/s; solar radiation = 800 W/m2 and 2nd. air temperature = 40.6°C; relative humidity = 30%; wind speed = 0.5 m/s; solar radiation = 0 W/m2) and two neutral environments: 20°C WBGT (1st: air temperature = 19.1°C; relative humidity = 30%; wind speed = 0.5 m/s; solar radiation = 800 W/m2 and 2nd. air temperature = 28.5°C; relative humidity = 30%; wind speed = 0.5 m/s; solar radiation = 0 W/m2], over an equal number of days. The aforementioned environmental scenarios were randomly allocated for each volunteer. To minimize participant bias, the true purpose of the study was hidden from the volunteers. Of course, once the data collection was completed, all volunteers were informed about the true purpose of the study and gave their permission to analyze and publish these data. During this blinded randomized controlled trial, all volunteers participated four times in an experimental protocol with a total duration of 03:20:00, following an hour of preparation and baseline tests. The protocol had three main time periods [rest (two hours), work (cycling) at 100 W (one hour), and recovery (twenty minutes)]. Anthropometrical data [age; body stature (Seca 213; seca GmbH & Co. KG; Hamburg, Germany); body mass (BC1000, Tanita corporation, Tokyo, Japan); body fat (DXA scan: Lunar DPX Madison, GE Healthcare, Wisconsin, USA); and lean mass (DXA scan: Lunar DPX Madison, GE Healthcare, Wisconsin, USA)] were collected two days prior to the experiments.

Volunteers were euhydrated prior to the experiments. Hydration status was assessed using a handheld refractometer (ATAGO Ltd, Tokyo, Japan) and determined as either euhydrated (USG < 1.020) or dehydrated (USG ≥ 1.020) according to the current guidelines. Water consumption was restricted during the experimental protocol. The same clothing consisting of a light-blue t-shirt (100% cotton), a black exercise short pant (100% polyester), and a pair of medium-high socks (100% cotton) were used by volunteers throughout the experiments. A pair of sunglasses was mandatory to be worn throughout the experiments. Furthermore, experiments took place during the same hour of the day for each participant and an 8-hour fasting was ensured prior to the experiments. Furthermore, participants were requested to avoid caffeine and alcohol consumption for at least twelve hours before the experiments, as well as to avoid salt and sugar consumption eight hours before the experiments.

During the study, continuous heart rate, core temperature, mean skin temperature, skin blood flow, and sweat rate were measured. Specifically, heart rate was collected using wireless heart rate monitors (Polar Team2. Polar Electro Oy, Kempele, Finland). Core temperature was collected using telemetric capsules (BodyCap, Caen, France). Skin temperature from four sites was measured using wireless thermistors (iButtons type DS1921H, Maxim/Dallas Semiconductor Corp., USA) and was expressed as mean skin temperature according to Ramanathan [mean skin temperature = 0.3(chest + arm) + 0.2(thigh + leg). Skin blood flow was measured with a laser Doppler flowmeter (PeriFlux 4000, Perimed, Stockholm, Sweden) at right forearm (brachioradialis) and leg (gastrocnemius). The probe (PROBE 413 Integrating Probe, Perimed, Stockhold, Sweden) was held in place with a plastic holder (PH 13, Perimed, Stockhold, Sweden). Sweat rate was measured at three regions [forehead, thigh (quadricep), and arm (bicep)] using ventilated capsule method. Thermal comfort (1 = comfortable; 5 = extremely uncomfortable), thermal sensation (-3 = cold; +3 = hot), and perceived exertion (6 = no exertion at all; 20 = maximal exertion), alongside cognitive performance (vigilance, divided attention, memory test, and reaction time) were assessed at baseline, pre work condition (01:40:00), and post work (03:00:00) conditions. Volunteers entered the chamber five minutes prior to the experiments to install data loggers and accompanied sensors on their body.

ELIGIBILITY:
Inclusion Criteria:

* Healthy non-smoker individuals who exercise at least three times per week

Exclusion Criteria:

* Non healthy individuals and smokers

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 7 (Actual)
Dates: Start 2019-02-15 (Actual); Primary Completion 2019-05-27 (Actual); Study Completion 2019-05-27 (Actual)

PRIMARY OUTCOMES:
Heart rate | 03 hours and 20 minutes
  Heart rate data were continuously monitored using a Polar Team system (Polar® Team 2, Polar Electro Oy, Kempele, Finland
Mean skin temperature | 03 hours and 20 minutes
  Temperature at the skin surface area was continuously monitored using iButton sensors (type DS1921 H, Maxim/Dallas Semiconductor Corp., USA)
Core body temperature | 03 hours and 20 minutes
  Core body temperature was assessed throughout the entire protocol using telemetric capsules (e-Celsius, BodyCap, Caen, France) that was given to the workers to ingest prior to their work shift
Skin blood flow | 03 hours and 20 minutes
  Skin blood flow was measured throughout the entire protocol with a laser Doppler flowmeter (PeriFlux 4000, Perimed, Stockholm, Sweden) at right forearm (brachioradialis) and leg (gastrocnemius)
Sweat rate | 03 hours and 20 minutes
  Sweat rate was measured throughout the entire protocol at three regions [forehead, thigh (quadricep), and arm (bicep)] using ventilated capsule method
Perceived exertion | Participants were assessed at baseline and every half an hour up until the end of the protocol at "hour 3".
  We used the Borg 20th Scale (6 = no exertion at all; 20 = maximal exertion)
Cognitive performance (Vigilance) | Participants were assessed at baseline, at 1 hour and 40 minutes, and at "hour 3".
  Vigilance was assessed via vigilance test. In this task two squares arranged vertically. A pattern jumps from one square to the other. Sometimes the pattern remains in one square. In this case volunteers had to touch the screen of a tablet computer as fast as possible. The total duration for the current task was set to 6 minutes. This is a well-known vigilance test described in the Test for Attentional Performance and previously used in the literature.
Thermal comfort | Participants were assessed at baseline and every half an hour up until the end of the protocol at "hour 3".
  Thermal comfort was assessed via the thermal comfort scale (1 = comfortable; 5 = extremely uncomfortable).
Thermal sensation | Participants were assessed at baseline and every half an hour up until the end of the protocol at "hour 3".
  Thermal sensation was assessed via the thermal sensation scale (-3 = cold; +3 = hot)
Cognitive performance (Divided Attention) | Participants were assessed at baseline, at 1 hour and 40 minutes, and at "hour 3".
  Divided attention task incorporates both auditory and visual stimuli in parallel. During the test a number of visual stimuli (crosses) appear in a random configuration in a 4X4 matrix. At the same time volunteers hear high and low beeps in a random order. The task is to detect whether crosses form a square and at the same time two high or low beeps are emitted twice in a row. This is a well-known vigilance test described in the Test for Attentional Performance and previously used in the literature.
Cognitive performance (Memory Test) | Participants were assessed at baseline, at 1 hour and 40 minutes, and at "hour 3".
  This is a computerized version of Sternberg's memory task. In this task volunteers had to observe carefully a random sequence of one to six digits (0 to 9) painted in white and displayed for 1.2 seconds each. Thereafter, a two second delay was followed by a random test digit filled in yellow color. Participants had to response as fast as possible by pressing "yes" or "no" button to indicate where the yellow digit appeared in the previous sequence or not, respectively. In this test participants were tested in 24 trials.
Cognitive performance (Reaction Time) | Participants were assessed at baseline, at 1 hour and 40 minutes, and at "hour 3".
  In this task participants had to respond as quickly as possible, by untouching the screen, after receiving a visual or acoustic stimulus.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Flouris, Principal Investigator — andreasflouris@gmail.com
Locations (1):
- FAME Lab, Department of Exercise Science, University of Thessaly, Trikala, Thessaly, Greece

IPD SHARING:
Plan to Share IPD: No